CLINICAL TRIAL: NCT06477328
Title: Treatment Compliance of Patients Diagnosed With Chronic Obstructive Pulmonary Disease And Their Quality of Life After Follow-up: Evaluation Via Telemedicine
Brief Title: Evaluating Chronic Obstructive Pulmonary Disease (COPD) Patients' Treatment Compliance and Quality of Life Via Telemedicine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Etlik City Hospital (Other Government)
Responsible Party: Principal Investigator, Zeynep Sena Doğan, MD, Gazi University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: GAZISOLMAZ01
Record Dates: First submitted 2024-06-17; First posted 2024-06-27 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: Telehealth; Copd
Keywords: telemedicine; copd; inhaler adherence; inhaler technique
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Telemedicine

STUDY DESIGN:
Intervention Model Description: It is a prospective, randomized controlled, method clinical research study. Patients who were hospitalized with COPD exacerbation in the last year were included in the study and were divided into 2 groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telemedicine group (Active Comparator): The study participants were evaluated through telemedicine visits at specific intervals after the baseline visit, with the following schedule:
  * 1st visit: At day 10 post-baseline
  * 2nd visit: At the end of the 1st month
  * 3rd visit: At the end of the 3rd month
  These visits were conducted by the principal investigator using telemedicine. Additional telemedicine visits were arranged for patients in the telemedicine group as required.
  Interventions: Procedure: Telemedicine
- Control group (No Intervention): The visits for the control group, due to being conducted face-to-face in the outpatient clinic, were carried out by the routine attending physician at the clinic, who was not aware of the study. As suggested in the discharge recommendations during the baseline visit (0th visit) for the control group, they were advised to return for a follow-up visit on the 10th day and to schedule these follow-up appointments through the hospital's system. No intervention was made to facilitate the scheduling of these appointments.

INTERVENTIONS:
Procedure: Telemedicine — Video calls were made with the telemedicine group.
  Arms: Telemedicine group

SUMMARY:
The Covid-19 pandemic has disrupted the follow-up and treatment processes for patients, and telemedicine has emerged as an important alternative method. Our aim was to test compare COPD Assessment Test (CAT) scores, inhaler treatment techniques and adherence between telemedicine-mediated healthcare and healthcare provided face-to-face.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were diagnosed with COPD according to Global Initiative for Obstructive Lung Disease (GOLD)
* GOLD spirometric grade 3-4
* At least one hospital admission in the past year
* Acceptable score on the Mini-Mental State Examination
* Residing in Ankara
* Patient or caregiver must understand the process and be able to provide clear information
* Medical records and laboratory test results must be accessible to healthcare professionals
* Patient must have access to prescribed medications
* Comorbidities outside of the lungs are included

Exclusion Criteria:

* Patients diagnosed with asthma
* Patients with lung cancer
* Patients with combined pulmonary fibrosis and emphysema
* Patients with active infections such as pneumonia or COVID-19
* Patients being followed for COPD without spirometry
* Patients with low cognitive function as determined by the Mini-Mental State Examination
* Patients who do not consent to participate in the study
* Patients lacking adequate social support
* Patients with COPD grade 1-2
* Patients with no hospital admissions in the past year
* Patients diagnosed with psychotic disorders
* Patients residing outside of Ankara
* Patients enrolled in inpatient or supervised outpatient rehabilitation programs
* Patients unable to use telemedicine devices or without a caregiver to assist
* Patients and caregivers having difficulty providing information
* Patients without internet access or video call capabilities at home

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-10-15 (Actual)

PRIMARY OUTCOMES:
Inhaler adherence | 3 months
  At the end of 3 months, inhaler adherence was compared. A 6-item Inhaler Adherence Scale (IAS) was used to evaluate inhaler treatment compliance. If the patient answered "yes" to even one of the items, they were deemed non-compliant.
  The questions:
  ''During the last 3 months;
  * have you at times been careless about using your inhaler or nebulizer?,
  * have you ever forgotten to use your inhaler or nebulizer?
  * have you ever stopped using your inhaler because you felt better?
  * have you ever stopped using your inhaler or nebulizer because you felt worse?
  * have you ever used your inhaler or nebulizer less than the doctor prescribed because you felt better?
  * have you ever used your inhaler or nebulizer more than the doctor prescribed because you felt you were having an attack?''.

SECONDARY OUTCOMES:
COPD Assesment Test (CAT) score | 3 months
  The aim of the investigator's study is to test whether telemedicine is a safe and effective method for the follow-up of patients with advanced-stage COPD after exacerbations, to see if there is a difference in treatment adherence after 3 months of observation compared to face-to-face healthcare services, and to evaluate if there is a difference in CAT scores.
  The COPD Assessment Test (CAT) is a questionnaire for people with COPD. It is designed to measure the impact of COPD on a person's life, and how this changes over time.
  Range of CAT scores from 0-40. Higher scores denote a more severe impact of COPD on a patient's life.

CONTACTS AND LOCATIONS:
Locations (1):
- Gazi University, Ankara, Turkey (Türkiye)

REFERENCES:
- [Derived] Dogan ZS, Kokturk N. Evaluation of patients diagnosed with chronic obstructive pulmonary disease in terms of treatment compliance and quality of life after follow-up with telemedicine: a randomized controlled trial. BMC Pulm Med. 2025 Aug 26;25(1):408. doi: 10.1186/s12890-025-03854-z. PMID 40859183